CLINICAL TRIAL: NCT07256470
Title: Salivary Replication of BK Virus in Post-kidney Transplant
Acronym: BKSAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PI2024_843_0093
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: BK Virus; Salivary Replication; Kidney Transplantation; Nephropathy; DNAemia
Keywords: BK virus; salivary replication; kidney transplantation; nephropathy; DNAemia
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Salivary self-collection — Salivary self-collection on the day of the kidney transplant then at 1, 3, 6, 9 and 12 months

SUMMARY:
BK virus infection in kidney transplantation can compromise graft function. Current data suggest that BK virus nephropathy results not only from transmission of virus from the donor but also from reactivation of latent virus in the recipient. However, no study has investigated the possibility of respiratory transmission. This study would provide a better understanding of the pathophysiology of BK virus infection in kidney transplant recipients. The investigators would study viral replication of BK virus in saliva, urine and blood of patients who received a kidney transplant at the Amiens University Hospital. For this, the investigators will collect salivary self-collection on the day of the kidney transplant then at 1, 3, 6, 9 and 12 months as well as a urine and blood sample. The investigators will measure BK viral load in these three samples at different times.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant recipients
* age ≥ 18 years

Exclusion Criteria:

* age < 18 years
* absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of BK positive saliva and blood samples | 12 months
  Compare the positivity of the BK virus viral load between the saliva sample and the urine and blood samples

SECONDARY OUTCOMES:
urinary BK virus concentration | 12 months
variation of BK virus genome | 12 months
  variation of BK virus genome in different samples
Immunoglobin concentrations | 12 months
  Immunoglobin concentrations in different samples

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No